CLINICAL TRIAL: NCT02785744
Title: Prevalence of Gaucher Among Patients With Osteopenia/Osteoporosis
Brief Title: Genzyme Osteopenia/Osteoporosis Study
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-00351
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving DEXA Scan: Gaucher patients referred for dual energy X-ray absorptiometry (DEXA scan), who were found to have T-score <-1.0.
  Interventions: Other: Gaucher disease DNA mutation analysis

INTERVENTIONS:
Other: Gaucher disease DNA mutation analysis

SUMMARY:
Gaucher disease is a most common genetic metabolic disease characterized by low platelet number, liver and spleen enlargement and various forms of bone diseases including low bone mineral density leading to brittle bones. Various treatment options are now available for this disease.

The purpose of this research study is to determine the prevalence of Gaucher disease in patients with low bone mineral density as observed by DEXA scan, which is a form of X-Ray of the bone.

DETAILED DESCRIPTION:
Gaucher disease is a potential secondary cause of low bone mineral density and it is prevalent among patients with low BMD. This cross sectional design study will measure point prevalence of Gaucher disease in patients with low bone mineral density (BMD).

ELIGIBILITY:
Inclusion Criteria:

* Patients > or equal to18 years and able to provide written consent.
* Patients who have had a bone density test demonstrating T-score <-1.0 on a DEXA scan within the past year or those who are prospectively referred for DEXA scan and who are later identified by their physician to have a DEXA T-score < -1.0.

Exclusion Criteria:

* Subject unable to read and sign consent form.
* Terminally ill subjects or subjects with serious co-morbidities (malignancy), which would limit the ability of the patient to participate in the study.
* Subjects with the following disorders or exposures
* Underlying skeletal dysplasia
* An endocrinologic/metabolic disease known to cause bone demineralization: including parathyroid dysfunction, hyperthyroidism, Cushing syndrome, hypogonadism, panhypopituitarism
* Cystic Fibrosis
* Exposure to medications that are known to cause low BMD including chemotherapy within past 2 years, chronic corticosteroid or phenytoin use within past 2 years
* Radiation exposure within the past 5 years
* Vitamin D deficiency is not an exclusion criteria as this is highly prevalent in the adult population under investigation as well as in patients with Gaucher disease. (9, 10)
* Subjects previously diagnosed with Gaucher Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in a cross-sectional design measuring point prevalence of Gaucher disease in patients with low bone mineral density. Low BMD is defined as T-Score <-1.0. In addition, prevalence stratified by age, gender, and menopausal status will be determined.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Population prevalence of Gaucher disease among patients with low bone mineral density | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Heather Lau, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States